CLINICAL TRIAL: NCT03759561
Title: A Prospective Randomized Trial on Comparison of Tracheal Intubation Using Videolaryngoscope Versus Fiberoptic Bronchoscope in Patients Undergoing Cervical Spine Surgery
Brief Title: Tracheal Intubation Using Videolaryngoscope vs Fiberoptic Bronchoscope in Patients With Cervical Immobilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VL_FOB
Record Dates: First submitted 2018-11-29; First posted 2018-11-30 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Intubation, Intratracheal
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Videolaryngoscope group (Active Comparator): In the videolaryngoscope group, tracheal intubation was performed using videolaryngoscope under cervical collar application.
  Interventions: Procedure: intubation with videolaryngoscope vs fiberoptic bronchoscope
- Fiberoptic bronchoscope group (Active Comparator): In the fiberoptic bronchoscope group, tracheal intubation was performed using fiberoptic bronchoscope via oral cavity under cervical collar application.
  Interventions: Procedure: intubation with videolaryngoscope vs fiberoptic bronchoscope

INTERVENTIONS:
Procedure: intubation with videolaryngoscope vs fiberoptic bronchoscope — Tracheal intubation was performed using either videolaryngoscope or fiberoptic bronchoscope under cervical collar application according to the group allocations

SUMMARY:
In patients with suspected cervical spine injury, cervical immobilization, such as manual in-line stabilization or cervical collar has been adopted to prevent further neurologic injury due to cervical motion. In these patients, tracheal intubation with direct laryngoscopy is often challenging due to limited mouth opening, neck flexion, and head extension. In this situation, videolaryngoscope and fiberoptic bronchoscope have been used for tracheal intubation in such patients. In this study, the initial success rate of tracheal intubation and intubation time between the videolaryngoscope and fiberoptic bronchoscope will be compared.

DETAILED DESCRIPTION:
Patients entered the operating room without premedication. Airway-related parameters (modified Mallampati score, interincisior gap, thyromental distance, sternomental distance, and retrognathia) were evaluated in the sitting position. After changing to the supine position, thyromental height was measured and patients were monitored with electrocardiography, pulse oximetry, non-invasive blood pressure measurement, and processed electroencephalography. Cotton towels were placed below the patient's head for horizontal alignment of the external auditory meatus and the suprasternal notch. After sufficient preoxygenation for > 3 min, total intravenous anaesthesia was induced using a target-controlled infusion of propofol and remifentanil (effect site concentration: 4 µg/mL for propofol and 4 ng/mL for remifentanil). After confirming loss of consciousness, rocuronium (0.6-0.8 mg/kg) was administered to facilitate tracheal intubation, and mask ventilation was conducted. During mask ventilation, its difficulty was assessed and the use of the oropharyngeal airway was recorded. For invasive blood pressure measurement, a 20-gauge catheter was placed on the patient's radial artery. Thereafter, the patient's head was placed in the neutral position and an cervical collar was applied to minimise neck movement during intubation.

About 90 s after administrating rocuronium, tracheal intubation was attempted by one of five attending anaesthesiologists with a collective history of more than 30 successful videolaryngoscopic and fiberscopic intubations. A reinforced tracheal tube was used in both groups. Orotracheal intubation was performed using a videolaryngoscope with a disposable Macintosh-typed blade and a malleable stylet in the videolaryngoscope group, and using a flexible fiberscope with an eyepiece in the fiberscope group. A tracheal tube was mounted on the stylet and flexible fiberscope in the videolaryngoscope and fiberscope groups, respectively. The stylet was angulated about 60° at the proximal margin of the cuff. Tracheal intubation was initially attempted without any assistance, including airway manoeuvres and devices. If additional airway manoeuvres including external laryngeal manipulation (ELM), jaw thrust, and tongue traction were required during intubation attempts, they were performed by an assistant and noted. After confirming the glottis, the percentage of glottic opening (POGO) score was recorded just before inserting the tracheal tube into the trachea. The tracheal tube was inserted into the trachea after removing the stylet and confirming the carina in the videolaryngoscope and fiberscope groups, respectively. Successful intubation was confirmed by waveform capnography. The time from oral insertion of the intubation device to obtainment of the glottis view (glottis visualisation time), to placement of the tracheal tube (tube placement time), and to detection of the waveform capnograph (capnograph detection time) were also measured.

A maximum of three intubation attempts were allowed for the same anaesthesiologist, with a 180-s time limit for each attempt. If the peripheral oxygen saturation (SpO2) decreased to below 90% during the intubation attempt, the attempt was considered to have failed, and rescue mask ventilation was conducted until SpO2 reached 100%. Cases where tracheal intubation was unsuccessful on all three attempts were recorded as intubation failure.

After surgery, intubation-related airway complications were investigated. Airway injuries (blood in the oral cavity, blood staining on the tracheal tube, gum bleeding, and dental trauma) were assessed at the end of surgery. In addition, hoarseness and sore throat were evaluated at 1 h and 24 h after surgery. The severity of sore throat was measured using a numeric rating scale (NRS; 0: no pain, 10: worst pain imaginable).

Mean blood pressure (MBP), heart rate (HR), SpO2, and bispectral index (BIS) were recorded just before the intubation attempt and at 1 min after successful intubation. Other perioperative data (demographic, anaesthetic, and surgical data) were collected from electronic medical records.

ELIGIBILITY:
Inclusion Criteria:

* Patients who require tracheal intubation
* Adult patients aged 20-80
* American Society of anesthesiologists physical status classification Ⅰ-Ⅲ

Exclusion Criteria:

* patient's refusal
* patients had a high risk of aspiration, history of gastroesophageal reflux disease, coagulopathy, previous history of radiation therapy on the neck and airway surgery, and upper airway lesions (i.e., tumor, polyp, inflammation, trauma, abscess, and foreign body)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
The initial success rate | intraoperatively
  The first-pass success was defined as successful tracheal intubation on a single attempt in all stages of tracheal intubation

SECONDARY OUTCOMES:
intubation time | intraoperatively
  Intubation time was defined as time interval between insertion of the device into the oral cavity and withdrawal of the device from the oral cavity.
the incidence of complication | intraoperatively to 1hour and 24 hours after the surgery
  The complications after the procedure included blood in the oral cavity, blood staining on the endotracheal tube, sore throat, and hoarseness. Blood in the oral cavity and blood staining on the endotracheal tube will be evaluated intraoperatively. Sore throat and hoarseness will be evaluated at 1 hour and 24 hours after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hee-pyoung Park, MD,PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No